CLINICAL TRIAL: NCT03876639
Title: Topical Application of Highly Concentrated Water-in-oil Emulsions: Physiological Skin Parameters and Skin Penetration in Vivo - A Pilot Study
Brief Title: Topical Application of Highly Concentrated Water-in-oil Emulsions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Lisa Binder, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SkinStudy 2019.1
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Skin Physiology; Dermal Administration; Emulsions
Keywords: Water-in-oil emulsion; Confocal Raman spectroscopy; Skin parameters; Tape stripping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPM_2/18 (Active Comparator): Application of formulation IPM_2/18
  Interventions: Other: Application of emulsion; Procedure: Measurement of physiological skin parameters; Procedure: Tape stripping
- PAR_2/18 (Active Comparator): Application of formulation PAR_2/18
  Interventions: Other: Application of emulsion; Procedure: Measurement of physiological skin parameters; Procedure: Tape stripping

INTERVENTIONS:
Other: Application of emulsion — Daily application of the assigned formulation on the non-dominant volar forearm for 4 weeks
Procedure: Measurement of physiological skin parameters — Weekly measurement of physiological skin parameters using confocal Raman spectroscopy, Corneometer® CM 825, Sebumeter®, Skin-pH-Meter®, AquaFlux® and Epsilon®
Procedure: Tape stripping — Removal of 40 adhesive strips after application of a model drug-loaded emulsion and determination of the transepidermal water loss

SUMMARY:
The purpose of this study is to I. determine the effect of repetitive application of newly developed silicone based formulations (placebo water-in-oil emulsions) on transepidermal water loss and other physiological skin parameters and II. investigate the skin penetration of the model drug fluorescein sodium in tape stripping studies to determine the in vivo penetration profile from the water-in-oil emulsions.

DETAILED DESCRIPTION:
Water-in-oil emulsions will be applied daily for a period of 4 weeks on the non-dominant volar forearm of voluntary participants. Several physiological skin parameters will be monitored in weekly intervals during the application period. Additional measurements will be carried out immediately before the start of the application and after a treatment-free recovery period of 2 weeks. The untreated forearm will be used as a reference.

Subsequent to the observational study, tape stripping experiments with fluorescein sodium-loaded formulations will be conducted on the non-dominant forearm of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent
* Female or male aged between 18 and 65 years

Exclusion Criteria:

* Pregnancy
* Chronic skin conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Change in transepidermal water loss | 6 weeks
  Influence of the application of the water-in-oil emulsions with different oil component - isopropyl myristate (IPM) or liquid paraffin (PAR) - on the transepidermal water loss (TEWL) using the AquaFlux Model AF200 Evaporimeter
Penetrated amount of fluorescein sodium into the skin using tape stripping/fluorescence spectroscopy | week 8
  Enhancement of the skin penetration of the model drug fluorescein sodium by the oil component isopropyl myristate in vivo using tape stripping combined with fluorescence spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided